CLINICAL TRIAL: NCT05652283
Title: An Exploratory Clinical Study of Neoadjuvant Therapy With Pamiparib Combined With Surufatinib for Advanced Ovarian Cancer: A Single-arm, Prospective, Single-center Clinical Study
Brief Title: Pamiparib Combined With Surufatinib for the Neoadjuvant Treatment of Unresectable Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bai-Rong Xia (Other)
Responsible Party: Sponsor-Investigator, Bai-Rong Xia, Chairman of Department of Gynaecology Surgery, Anhui Provincial Cancer Hospital
Organization: Anhui Provincial Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnhuiCancer
Record Dates: First submitted 2022-11-27; First posted 2022-12-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pamiparib; surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experience group (Experimental): Pamiparib 40 mg, BID, oral, 3 weeks as a cycle, 3 cycles Surufatinib 250 mg, QD, oral, 3 weeks as a cycle, 2 cycles
  Interventions: Drug: Pamiparib; Drug: Surufatinib

INTERVENTIONS:
Drug: Pamiparib — Pamiparib capsule 40 mg/time, twice a day, oral, 3 weeks as a cycle, 3 cycles
  Other Names: BAIHUIZE
Drug: Surufatinib — Surufatinib 250 mg/time, once a day, oral, 3 weeks as a cycle, 2 cycles
  Other Names: SULANDA

SUMMARY:
The goal of this type of clinical trial study is to evaluate the safety and efficacy of Pamiparib combined with Surufatinib as a new neoadjuvant therapy in newly diagnosed patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
Patients will have tests and exams to see if they are eligible for the clinical trial. If found eligible, the patient will receive Pamiparib twice daily and Surufatinib once daily taken by mouth every 3 weeks.

Patients who had no progression after neoadjuvant therapy were treated with surgery, and 4 cycles of chemotherapy were given after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Before any procedure of the test is started, informed consent must be provided and filed in the research center.
* Female subjects ≥ 18 years of age.
* Biopsy obtained by open surgery, laparoscopic surgery or thick needle puncture, pathologically confirmed as high-grade serous or endometrioid ovarian cancer, peritoneal cancer, or fallopian tube cancer (hereinafter referred to as ovarian cancer), FIGO stage III-IV.
* Detect tissue samples or blood samples through a testing agency designated by the research center to determine the HRR-related gene mutation or HRD mutation status of patients.
* The blood and tissue samples of patients before, during, and after treatment can be obtained, and the subjects agree to submit the blood and tissue samples to the Center for the expanded research purpose of the trial, such as possible gene-related research or tumor marker related research.
* At least one lesion can be measured by CT/MRI.
* The professional gynecological oncologists appointed by each center should judge the patients who can not achieve R0 tumor reduction or can not tolerate surgery.
* The criteria for failure to achieve R0 tumor reduction include but are not limited to:Fagotti endoscopic score ≥ 8 points；When the laparoscopic evaluation method is difficult to implement, the upper abdomen CT score can be ≥ 3 points;
* The judgment criteria of intolerable surgery can consider:Body mass index: BMI ≥ 40.0；Multiple chronic diseases；Malnutrition or hypoproteinemia Moderate to massive ascites；Newly diagnosed venous thromboembolism (except intermuscular venous thrombosis) (survival time greater than 12 weeks).
* Expected survival time > 12 weeks.
* The patient's ECOG score is 0-2.
* Good organ function, including:Bone marrow function: neutrophil count ≥ 1500/µ L; Platelet ≥ 100000/µ L; Hemoglobin ≥ 10g/dL；Liver function: total bilirubin ≤ 1.5 times the upper limit of normal value or direct bilirubin ≤ 1.0 times the upper limit of normal value; AST and ALT ≤ 2.5 times the upper limit of normal value, and when liver metastasis exists, it must be ≤ 5 times the upper limit of normal value Renal function: serum creatinine ≤ 1.5 times the upper limit of normal value, or creatinine clearance rate ≥ 60mL/min (calculated according to Cockcroft Gault formula).
* For women with fertility potential, the blood test or urine pregnancy test was negative within one week before enrollment. After enrollment, effective contraceptive measures must be taken, such as using physical barrier contraceptive methods (condoms) or complete abstinence; Oral, injectable, or implanted hormonal contraceptives are not allowed.

Exclusion Criteria:

* Personnel involved in the formulation or implementation of the research plan.
* Use other experimental research drugs and participate in other clinical drug experiments while the study is being conducted.
* At the same time of the study, use other new adjuvant therapies for tumors, including but not limited to chemotherapy, radiotherapy, immunotherapy, microbial therapy, traditional Chinese medicine, and other experimental therapies.
* People who are known to be allergic to active or inactive ingredients of Pamiparib, Surufatinib or drugs with similar chemical structures to the two drugs.
* Unable to swallow the oral drug, and suffering from any gastrointestinal disease that may interfere with the absorption and metabolism of the study drug, such as uncontrollable nausea and vomiting, gastrointestinal obstruction or malabsorption.
* Have received any anti-cancer treatment related to ovarian cancer.
* Have received known or possible PARP inhibitor treatment in the past.
* Symptomatic or uncontrolled brain metastasis requiring simultaneous treatment, including but not limited to surgery, radiation and/or corticosteroids, or clinical manifestations of spinal cord compression.
* Major surgery was performed within 3 weeks before the start of the study, or it has not recovered after surgery.
* Subjects had other malignant diseases in the past 3 years, except for effectively treated skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ or cervical carcinoma in situ.
* The patient has myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) previously or currently diagnosed.
* Suffering from serious and uncontrollable diseases or the investigator judged that the subject was generally not suitable for the study, including but not limited to: active virus infection, such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.; Severe cardiovascular disease, uncontrollable ventricular arrhythmia, and myocardial infarction in the last 3 months; Uncontrolled seizures, unstable spinal cord compression, superior vena cava syndrome or other mental disorders that affect the patient's informed consent; Hypertension beyond drug control; Immune deficiency (excluding splenectomy) or other diseases that the researchers believe may expose the patient to high-risk toxicity.
* Any medical history or existing clinical evidence indicates that there may be circumstances that may confuse the study results, interfere with patients' compliance with the trial protocol during the whole study treatment period or are not in the best interests of patients.
* The patient received platelet or red blood cell infusion within 3 days before the start of treatment of the study drug.
* Patients who are pregnant or nursing, or who are expected to become pregnant during the study treatment.
* There are unresolved previous treatment toxicity (≥ grade 2, excluding alopecia, neuralgia, lymphocytopenia, and depigmentation of skin) in clinic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3-month
  the percentage of patients received R0 resection after Pamiparib combined with Surufatinib neoadjuvant therapy

SECONDARY OUTCOMES:
Overall Response Rate (ORR) After Neoadjuvant treatment | 3-month
  Overall Response Rate according to RECIST1.1 after Neoadjuvant treatment. ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions.
Pathological complete remission rate | 3-month
  No residual invasive carcinoma was found under the microscope, but ductal carcinoma in situ could be found; In addition, compare the amount of cancer cells in the specimen before and after the new adjuvant therapy, and use of the Miller Payne grading system to evaluate the effect of the new adjuvant therapy
12-month disease-free survival rate | 12 months
  The rate of patients who did not have any event from the beginning of enrollment to 12 months, including disease progression, inoperable, local or remote recurrence, and death from any cause
12-month survival rate | 12 months
  Rate of patients who did not have a death event from enrollment to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Rong Xia, MD, Study Chair — Anhui Provincial Cancer Hospital; Wenjing Jiang, Study Director — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China